CLINICAL TRIAL: NCT01900119
Title: A Description of the Oral Microbiome of Patients With Severe Aplastic Anemia
Brief Title: A Description of Bacteria in the Mouths of Patients With Severe Aplastic Anemia
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 130161; 13-CC-0161
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-09-23

CONDITIONS: Severe Aplastic Anemia (SAA)
Keywords: Oral Microbiome; Next Generation Sequencing
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- This research is being done to describe the types of bacteria found in the mouths of patients who have severe aplastic anemia (SAA) and are treated with drugs that suppress the immune system or with stem cell transplant. People with SAA who receive these treatments are more likely to get infections. Studies show that there might be a link between the bacteria in your mouth and those bacteria that can cause infections. The bacteria found in the mouths of patients with SAA will be described.

Objectives:

- To understand the changes in mouth bacteria that are related to treatment and to describe the oral bacterial environment.

Eligibility:

* Adults at least 18 years of age who are going to be treated for SAA.
* Healthy volunteers at least 18 years of age.

Design:

* Participants will answer questions about their medical history and dental care. Their mouths will be examined.
* Participants with SAA will be tested during treatment for their disease, over the course of 1 year. All participants with SAA will be tested at 3 scheduled appointments. Any participants who require a breathing tube will receive additional tests.
* Healthy volunteers will be tested during 1 visit.
* Participants will give two samples each time. A saliva sample will be taken with a disposable padded tool. Skin cells will be collected from the tongue with a small plastic brush.

DETAILED DESCRIPTION:
The mouth is a complex biological ecosystem normally containing over 700 different species of bacteria. Some of these bacteria live in an exopolysacchride matrix biofilm and occupy specific niches in this complex oral environment. Understanding the oral environment and the microbiota that inhabit it will assist in determining their impact on health and disease. There are several studies in critically ill patients demonstrating changes in oral bacteria related to acute illness. Identification of respiratory pathogens in the mouth has led researchers to hypothesize that a relationship exists between the oral cavity and pulmonary infections. This descriptive study will characterize the oral microbiota of patients who have severe aplastic anemia (SAA). Patients will be followed for 1 year after treatment for development of respiratory symptoms that require intubation. A difference in the oral microbiome will be identified in specimens collected before and after treatment.

ELIGIBILITY:
* All adult patients who are scheduled to receive treatment for SAA will be screened for this protocol. These patients will be recruited from the numerous protocols that are actively accepting new research participants at the Clinical Center, NIH.

INCLUSION CRITERIA

Any adult patient (greater than or equal to18 years of age), diagnosed with SAA.

EXCLUSION CRITERIA

Any SAA patient found to have significant tooth loss from decay or is edentulous are excluded. This exclusion criteria will be assessed by the PI or her representative prior to signing the informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12-12; Primary Completion 2016-07-05 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Compare the oral microbiome of SAA patients prior to treatment and after treatment. | one year following enrollment
  Change in the oral microbiome of patients with SAA. Bacterial data obtained from sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ames, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Socransky SS, Haffajee AD. Periodontal microbial ecology. Periodontol 2000. 2005;38:135-87. doi: 10.1111/j.1600-0757.2005.00107.x. No abstract available. PMID 15853940
- [Background] Mager DL, Ximenez-Fyvie LA, Haffajee AD, Socransky SS. Distribution of selected bacterial species on intraoral surfaces. J Clin Periodontol. 2003 Jul;30(7):644-54. doi: 10.1034/j.1600-051x.2003.00376.x. PMID 12834503
- [Background] Kolenbrander PE, Andersen RN, Blehert DS, Egland PG, Foster JS, Palmer RJ Jr. Communication among oral bacteria. Microbiol Mol Biol Rev. 2002 Sep;66(3):486-505, table of contents. doi: 10.1128/MMBR.66.3.486-505.2002. PMID 12209001